CLINICAL TRIAL: NCT02382835
Title: Metal-on-metal Hip Prostheses: Do They Have Systemic Effects?
Acronym: HipLink
Status: Completed | Type: Observational
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Professor Alister Hart, Professor of Orthopaedics, Royal National Orthopaedic Hospital NHS Trust
Other Study IDs: 1
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Hip Replacement; Heart Failure
Keywords: metal-on-metal
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metal-on-Metal Hip Replacement
- Other Hip Replacement: Other types of hip replacement, such as metal-on-polyethylene or ceramic-on-ceramic

SUMMARY:
This study aims to determine whether subjects who underwent large-diameter metal-on-metal hip arthroplasty are more likely to have developed heart failure or other conditions as compared to subjects with conventional hip replacements.

We plan to link the National Joint Registry for England, Wales and Northern Ireland to the National Heart Failure Audit and GP records.

DETAILED DESCRIPTION:
Background: Chronic systemic exposure to very high concentrations of cobalt or chromium following large diameter metal-on-metal hip resurfacing or hip replacement (MOMHR) associates with cardiac, thyroid, visual, hearing, and peripheral neurological deficits. Chronic exposure to lower circulating metal levels also associates with changes in cardiac function and bone metabolism in case-control analyses. However, it remains unclear what the risk of these problems is in the general population exposed to MOMHR.

Aims: We aim to establish the prevalence of cardiac, endocrine, neurological disorders, and distant site fracture history (forearm, spine) in recipients of MOMHR, and establish whether this differs to that found in the general population of the same age and sex distribution, and also to recipients of hip replacement using a conventional bearing.

Methods: We will use NJR data linked to the Clinical Practice Research Dataset (CPRD) to establish the prevalence of cardiac, endocrine, neurological disorders, and distant site fracture history (forearm, spine) in the 3 study populations.

Outcome measures: All defined as the event occurring at any point following MOMHR surgery.

Primary outcome measure:

History of cardiac failure, as defined by IDC9-CM code 150, or equivalent CPRD codes

Secondary outcome measures:

1. History of treated or untreated acquired hypothyroidism (ICD9 244.8), or equivalent
2. Fracture history at a site distant to the ipsilateral hip (ICD9 820.00 to 826.1)
3. Acquired neurological disorders, including extra-pyramidal disorders (ICD9 332 and 333), spinocerebellar degenerative disease (ICD9 334) and other paralytic syndromes (ICD9 344)
4. Acquired blindness and low vision (ICD9 369)
5. Acquired hearing loss (ICD9 389)

Analyses will be conducted with age, sex, and joint disease diagnosis matching. Analyses will be stratified by sex to establish whether any differences are sex specific, and adjusted for age and other comorbidities, including history of type 2 diabetes, pre-existing ischaemic heart disease, hypertension, and pre-existing use of drugs that may affect cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable patients registered with an up to standard practice which participates in the CPRD linkage scheme.
* Have at least 6 (or 12) months of valid follow up in the primary care database.
* Primary or revision hip replacement on National Joint Registry (NJR) database occurring to during the period of availability of metal-on-metal implants, and during the available primary care follow up period for that patient.
* NHS number and other linkage identifiers available for both data sources
* Patient consent to NJR use of patient data (which is present for 99.6% of records on NJR)

Exclusion Criteria:

* Procedures on NJR database performed in Wales, Scotland and Northern Ireland (as these areas are not been included in the CPRD linkage scheme)
* Patients whose hips were implanted in the past 6 months - this exclusion criterion will be implemented post linkage of the data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Description= Patients with a total hip replacement on the National Joint Registry that can be linked to either National Institute for Cardiovascular Outcomes Research (NICOR) or the Clinical Practice Research Datalink (CPRD) Geography = England Setting= Primary, Secondary and Tertiary care Dates = 1st April 2003 (the start of data collection for the National Joint Registry) to present
Sampling Method: Probability Sample
Enrollment: 800000 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Heart failure | 6 months onwards

SECONDARY OUTCOMES:
History of treated or untreated acquired hypothyroidism or equivalent | 6 months onwards
Fracture history at a site distant to the ipsilateral hip | 6 months onwards
Acquired neurological disorders, including extra-pyramidal disorders spinocerebellar degenerative disease and other paralytic syndromes | 6 months onwards
Acquired blindness and low vision | 6 months onwards
Acquired hearing loss | 6 months onwards

CONTACTS AND LOCATIONS:
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, United Kingdom